CLINICAL TRIAL: NCT02405325
Title: PEP4PA - Peer Empowerment Program for Physical Activity in Low Income and Minority Seniors
Brief Title: Peer Empowerment Program for Physical Activity in Low Income and Minority Seniors
Acronym: PEP4PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Loki Natarajan, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 150336; R01HL125405 (NIH)
Record Dates: First submitted 2015-03-20; First posted 2015-04-01 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Physical Activity
Keywords: physical activity; multilevel; cost-effectiveness; older adults
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): The program will be run by peer Leaders and senior center staff with the support of UCSD staff. Participants will work towards a 2000 increase in daily steps through self-paced incidental walking and peer led group walks.
  Interventions: Behavioral: Physical Activity
- Usual Care (No Intervention): Measurement at baseline, 6, 12, 18 and 24 months only with a health related event at each time point.

INTERVENTIONS:
Behavioral: Physical Activity — intervention activities will remain at the daily level, including using pedometers, having daily goals, attendance at Peer lead group walks and recognition of efforts through monthly celebrations and bi-weekly goal tracking with peer Health Coaches.
  Arms: Physical Activity

SUMMARY:
Older adults are the least active population group in the US. Yet, research has shown that an increase in physical activity (PA) can have immediate and profound effects on cardiovascular health. Older adults who are active use significantly fewer health care resources, and with the increasing number of older adults in the US it is imperative to curb health care expenditure in this group. PEP4PA (Peer Empowerment Program 4 Physical Activity) is a multilevel intervention aimed at increasing physical activity levels in a population of low income and ethnically diverse older adults. It will be delivered in centers by trained older adults. Participants will work towards a daily increase of 2000 steps per day through self-paced incidental walking, peer led group walks, and attendance at existing center PA classes. They will also work on projects to increase opportunities to be physically active at their center or in the surrounding neighborhood.

DETAILED DESCRIPTION:
In a 2-year cluster randomized controlled field trial of 408 ethnically diverse, older adults (50+ years old) in 12 low income community centers serving seniors in San Diego County the investigators will investigate:

1. The efficacy of PEP4PA (Peer Empowerment Program 4 Physical Activity) to reduce disparities in PA by increasing the percentage of participants achieving 150 minutes of PA per week at 6 and 12 months. Hypothesis: Participants in PEP4PA will significantly increase PA minutes in moderate intensity (measured objectively by accelerometry) to a greater extent than older adults receiving usual care (e.g. normal PA programing) in control centers and a greater percent will meet NHANES criteria for weekly PA.
2. The efficacy of PEP4PA to improve physical functioning, blood pressure (BP), depressive symptoms and quality of life. Hypothesis: Participants in PEP4PA will significantly increase their physical functioning (measured objectively by the short physical performance battery and 6 minute timed walk), decrease their systolic BP (mmHg) and reporting of depressive symptoms, and improve their quality of life scores (measured at baseline, 6 & 12 months) to a greater extent than older adults in control centers.
3. Assess the incremental cost effectiveness ratio (ICER) of PEP4PA in terms of cost per MET hour and cost per QALY compared to usual programming in the control centers at 12 months.
4. Evaluate the impact of PEP4PA on secondary outcomes such as sedentary time and sleep quality (measured by accelerometry), cognitive/executive functioning, and walking routes (from GPS) at 12 months.

Exploratory aims: 5. Examine individual, interpersonal, organizational, and environmental factors that affect implementation & behavior change. 6. Assess the efficacy, effectiveness and ICER of PEP4PA at 24 months

ELIGIBILITY:
Inclusion Criteria:

* are 50 years or older
* have not had a fall that resulted in a hospitalization in the past 12 months
* able to complete a 3 meter walking test within 30 seconds
* able to read and write in English
* able to walk without assistance from another person
* able to wear study devices and complete assessments
* able to complete written surveys without assistance
* able to attend regular study activities at the center
* able to provide written informed consent and complete a post consent comprehension assessment
* able to commit approximately 10 hours per week to study activities (peer Health Coach only)
* active for 20 minutes per day on at least 3 days per week (peer Health Coach only)

Exclusion Criteria:

1. are younger than 50 years,
2. have had a fall that resulted in a hospitalization in the last 12 months,
3. cannot complete the walking test within 30 seconds,
4. are not able to read and write in English,
5. cannot walk without human assistance
6. unable to wear study devices and complete assessments,
7. unable to complete written surveys without assistance,
8. cannot regularly attend study activities at the center,
9. are not able to provide written informed consent,
10. do not adequately answer questions on the post consent test,
11. Participated in the Community of Mine research study (UCSD)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Rich P, Aarons GA, Takemoto M, Cardenas V, Crist K, Bolling K, Lewars B, Sweet CC, Natarajan L, Shi Y, Full KM, Johnson E, Rosenberg DE, Whitt-Glover M, Marcus B, Kerr J. Implementation-effectiveness trial of an ecological intervention for physical activity in ethnically diverse low income senior centers. BMC Public Health. 2017 Jul 18;18(1):29. doi: 10.1186/s12889-017-4584-1. PMID 28720079
- [Derived] Crist K, Full KM, Linke S, Tuz-Zahra F, Bolling K, Lewars B, Liu C, Shi Y, Rosenberg D, Jankowska M, Benmarhnia T, Natarajan L. Health effects and cost-effectiveness of a multilevel physical activity intervention in low-income older adults; results from the PEP4PA cluster randomized controlled trial. Int J Behav Nutr Phys Act. 2022 Jun 27;19(1):75. doi: 10.1186/s12966-022-01309-w. PMID 35761363

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity | Usual Care
Started | 267 | 209
Completed | 203 | 175
Not Completed | 64 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity | Usual Care | Total
Number analyzed (Participants) | 267 | 209 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (8.8) | 71.5 (9.1) | 71 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 144 | 359
  Male | 52 | 65 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 120 | 177 | 297
  Black or African American Black or African American | 113 | 4 | 117
  Asian | 6 | 15 | 21
  Other | 28 | 13 | 41
  Hispanic | 47 | 25 | 72
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 267 | 209 | 476

OUTCOME MEASURES:

1. Primary Outcome: Minutes of Physical Activity as Measured by Accelerometer
Description: Change in minutes of MVPA
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Physical Activity | Usual Care
Number analyzed (Participants) | 267 | 209
Minutes | 20.0 [16.1 to 23.9] | 19.2 [15.5 to 23.0]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Non-SAEs were not collected in a way that they can be separated.
Arm/Group | Physical Activity | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/267 | 0/209
Serious Adverse Events (participants affected / at risk) | 85/267 | 41/209
Other Adverse Events (participants affected / at risk) | 149/267 | 61/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=267) | Usual Care (N=209)
Serious physical injury (General disorders) | 10 (11) | 5 (5)
Fall (General disorders) | 21 (26) | 8 (8)
Prolonged hospitalization for any reason (General disorders) | 54 (71) | 28 (36)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=267) | Usual Care (N=209)
Other adverse event (General disorders) | 149 (311) | 61 (131) — Included reports of muscle cramping, joint pain, respiratory issues, infectious disease (i.e. flu) and chronic conditions, etc. for any reason, not related to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02405325/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02405325/SAP_001.pdf